CLINICAL TRIAL: NCT05124847
Title: Time Restricted Eating as a Treatment for Pediatric Obesity
Brief Title: TREating Pediatric Obesity
Acronym: TREPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: TREPO
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2021-10

CONDITIONS: Infant Obesity; Hepatic Steatosis; Metabolic Syndrome; Insulin Resistance; Dyslipidemias
MeSH Terms: conditions — Pediatric Obesity; Fatty Liver; Metabolic Syndrome; Insulin Resistance; Dyslipidemias | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRE-Control (Experimental)
  Interventions: Behavioral: Standard Care; Behavioral: Time restricted eating
- Control-TRE (Experimental)
  Interventions: Behavioral: Standard Care; Behavioral: Time restricted eating

INTERVENTIONS:
Behavioral: Standard Care — Participants will receive nutritional education sessions and will be instructed to maintain an intake window of at least 13 hours a day, preferably every day of the week and in any case at least 6 days a week.
Behavioral: Time restricted eating — A personalized progression will be established to progressively reduce the intake window during the first 10 days of intervention. After these first 10 days, the participants will be prescribed to limit food intake to a maximum of 10 hours a day, at least 5 days a week. Participant can freely select the time of day to place the intake window. However, it will be recommended to avoid making the last intake in the 3 hours before going to bed. After 4 weeks of intervention, the dietitian will invite them to reduce the intake window to 9 or 8 hours, if they consider it feasible, maintaining this new intake window during the last 4 weeks of intervention. The intake window can be maintained at 10 hours until the end of the study.

SUMMARY:
The main aim of the study is to collect preliminary information on the feasibility and efficacy of a time restricted eating intervention in Spanish children and adolescents with obesity and metabolic comorbidities. Two 8-week interventions will performed in a randomized crossover controlled design: a) reduction of the habitual eating window; b) standard care. Different measurements of body composition and cardiometabolic health markers will be performed along those weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 10 and 15 at the start of the study.
2. Obesity defined according to the criteria of the World Health Organization (BMI≥p95) and at least one of the following conditions:

   2.1. Hepatic steatosis confirmed by abdominal ultrasound in the previous 12 months.

   2.2. Triglycerides> 150 mg/dl, confirmed in analytical determination in the 4 weeks prior to the start of the study.

   2.3. HDL cholesterol <40 mg/dl, confirmed in analytical determination in the 4 weeks prior to the start of the study.

   2.4. LDL cholesterol> 135 mg/dl, confirmed in analytical determination in the 4 weeks prior to the start of the study.

   2.5. Insulin resistance, determined by elevated HOMA-IR confirmed by analytical determination in the 4 weeks prior to the start of the study.
3. Habitual eating window equal to or greater than 13 hours, with a response rate greater than 85%. Habitual eating window will be determined by self-registration during the screening process. Participants must properly record the habitual eating window in at least 12 of the 14 days that self-registration will be requested, and it must be equal to or greather than 13 hours at least 6 days a week.
4. Reporting to have maintained a stable weight and height status during the last two months (changes of less than 2 points in BMI (kg / m2)).
5. Agreement to participate in all phases and procedures of the study.

Exclusion Criteria:

1. Being diagnosed with an endocrine disorder, for example, diabetes mellitus under treatment with insulin or oral antidiabetics, thyroid disease, hypercortisolism, congenital adrenal hyperplasia.
2. Being diagnosed with a chronic digestive, rheumatological, neurological, cardiological, pneumological, autoimmune or infectious disease that affects energy metabolism.
3. Having undergone a surgical procedure that chronically alternates digestive or metabolic function.
4. Hypercholesterolemia requiring pharmacological treatment according to the Expert Consensus of the European Society of Arteriosclerosis specific to children.
5. Serum triglyceride concentration> 500 mg/dl.
6. Systolic or diastolic blood pressure values equal to or greater than the specific 95th percentile for age, sixth, and height, on 3 different occasions [42].
7. Hypertransaminasemia> 200 IU / L (5 times higher than the upper normal value in the laboratory), which would make it necessary to rule out other causes of liver disease.
8. Being diagnosed with an eating disorder or being at risk of developing these disorders, determined using the SCOFF questionnaire (two or more questions answered positively).
9. Presenting neurological alterations or chromosomopathies.
10. Consuming drugs or supplements that are likely to alter energy metabolism.
11. Being participating in a nutritional intervention or treatment of any kind, or having done so during the previous 3 months.
12. Having a demonstrable personal or professional relationship with any of the members of the investigation team.
13. Any other condition that in the opinion of the research team would contraindicate their participation.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Length of eating window | From week 0 to week 8
Body weight | week 8
Body fat mass | week 8
Lipid profile | week 8
HOMA-IR | week 8
Hepatic steatosis | week 8
Carotid intima-media thickness | week 8
Continuous glucose monitoring | From week 6 to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martín Masot, MD PhD, Principal Investigator — Hospital Regional Universitario de Málaga. Hospital Materno-Infantil.
Locations (1):
- Hospital Regional Universitario de Málaga. Hospital Materno-Infantil., Málaga, Spain

REFERENCES:
- [Background] Freedman DS, Sherry B. The validity of BMI as an indicator of body fatness and risk among children. Pediatrics. 2009 Sep;124 Suppl 1:S23-34. doi: 10.1542/peds.2008-3586E. PMID 19720664
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Gregg EW, Shaw JE. Global Health Effects of Overweight and Obesity. N Engl J Med. 2017 Jul 6;377(1):80-81. doi: 10.1056/NEJMe1706095. Epub 2017 Jun 12. No abstract available. PMID 28604226
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Background] Swinburn BA, Sacks G, Hall KD, McPherson K, Finegood DT, Moodie ML, Gortmaker SL. The global obesity pandemic: shaped by global drivers and local environments. Lancet. 2011 Aug 27;378(9793):804-14. doi: 10.1016/S0140-6736(11)60813-1. PMID 21872749
- [Background] Albaladejo-Vicente R, Villanueva-Orbaiz R, Carabantes-Alarcon D, Santos-Sancho J, Jimenez-Garcia R, Regidor E. Reversal of the Upward Trend of Obesity in Boys, but Not in Girls, in Spain. Int J Environ Res Public Health. 2021 Feb 14;18(4):1842. doi: 10.3390/ijerph18041842. PMID 33672817
- [Background] Geserick M, Vogel M, Gausche R, Lipek T, Spielau U, Keller E, Pfaffle R, Kiess W, Korner A. Acceleration of BMI in Early Childhood and Risk of Sustained Obesity. N Engl J Med. 2018 Oct 4;379(14):1303-1312. doi: 10.1056/NEJMoa1803527. PMID 30281992
- [Background] Perng W, Hajj H, Belfort MB, Rifas-Shiman SL, Kramer MS, Gillman MW, Oken E. Birth Size, Early Life Weight Gain, and Midchildhood Cardiometabolic Health. J Pediatr. 2016 Jun;173:122-130.e1. doi: 10.1016/j.jpeds.2016.02.053. Epub 2016 Mar 16. PMID 26995700
- [Background] Armstrong S, Li JS, Skinner AC. Flattening the (BMI) Curve: Timing of Child Obesity Onset and Cardiovascular Risk. Pediatrics. 2020 Aug;146(2):e20201353. doi: 10.1542/peds.2020-1353. Epub 2020 Jul 6. No abstract available. PMID 32632022
- [Background] Andes LJ, Cheng YJ, Rolka DB, Gregg EW, Imperatore G. Prevalence of Prediabetes Among Adolescents and Young Adults in the United States, 2005-2016. JAMA Pediatr. 2020 Feb 1;174(2):e194498. doi: 10.1001/jamapediatrics.2019.4498. Epub 2020 Feb 3. PMID 31790544
- [Background] Hartman C, Rennert HS, Rennert G, Elenberg Y, Zuckerman E. Prevalence of elevated liver enzymes and comorbidities in children and adolescents with overweight and obesity. Acta Paediatr. 2021 Mar;110(3):985-992. doi: 10.1111/apa.15469. Epub 2020 Jul 28. PMID 32649794
- [Background] Lycett K, Juonala M, Magnussen CG, Norrish D, Mensah FK, Liu R, Clifford SA, Carlin JB, Olds T, Saffery R, Kerr JA, Ranganathan S, Baur LA, Sabin MA, Cheung M, Dwyer T, Liu M, Burgner D, Wake M. Body Mass Index From Early to Late Childhood and Cardiometabolic Measurements at 11 to 12 Years. Pediatrics. 2020 Aug;146(2):e20193666. doi: 10.1542/peds.2019-3666. Epub 2020 Jul 6. PMID 32632021
- [Background] Spear BA, Barlow SE, Ervin C, Ludwig DS, Saelens BE, Schetzina KE, Taveras EM. Recommendations for treatment of child and adolescent overweight and obesity. Pediatrics. 2007 Dec;120 Suppl 4:S254-88. doi: 10.1542/peds.2007-2329F. PMID 18055654
- [Background] Styne DM, Arslanian SA, Connor EL, Farooqi IS, Murad MH, Silverstein JH, Yanovski JA. Pediatric Obesity-Assessment, Treatment, and Prevention: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2017 Mar 1;102(3):709-757. doi: 10.1210/jc.2016-2573. PMID 28359099
- [Background] Wilfley DE, Tibbs TL, Van Buren DJ, Reach KP, Walker MS, Epstein LH. Lifestyle interventions in the treatment of childhood overweight: a meta-analytic review of randomized controlled trials. Health Psychol. 2007 Sep;26(5):521-32. doi: 10.1037/0278-6133.26.5.521. PMID 17845100
- [Background] Viner RM, Hsia Y, Tomsic T, Wong IC. Efficacy and safety of anti-obesity drugs in children and adolescents: systematic review and meta-analysis. Obes Rev. 2010 Aug;11(8):593-602. doi: 10.1111/j.1467-789X.2009.00651.x. Epub 2009 Nov 17. PMID 19922432
- [Background] Hawley JA, Sassone-Corsi P, Zierath JR. Chrono-nutrition for the prevention and treatment of obesity and type 2 diabetes: from mice to men. Diabetologia. 2020 Nov;63(11):2253-2259. doi: 10.1007/s00125-020-05238-w. Epub 2020 Aug 6. PMID 32761356
- [Background] Di Francesco A, Di Germanio C, Bernier M, de Cabo R. A time to fast. Science. 2018 Nov 16;362(6416):770-775. doi: 10.1126/science.aau2095. PMID 30442801
- [Background] Aucouturier J, Duche P, Timmons BW. Metabolic flexibility and obesity in children and youth. Obes Rev. 2011 May;12(5):e44-53. doi: 10.1111/j.1467-789X.2010.00812.x. Epub 2010 Oct 26. PMID 20977601
- [Background] de Cabo R, Mattson MP. Effects of Intermittent Fasting on Health, Aging, and Disease. N Engl J Med. 2019 Dec 26;381(26):2541-2551. doi: 10.1056/NEJMra1905136. No abstract available. PMID 31881139
- [Background] Hutchison AT, Liu B, Wood RE, Vincent AD, Thompson CH, O'Callaghan NJ, Wittert GA, Heilbronn LK. Effects of Intermittent Versus Continuous Energy Intakes on Insulin Sensitivity and Metabolic Risk in Women with Overweight. Obesity (Silver Spring). 2019 Jan;27(1):50-58. doi: 10.1002/oby.22345. PMID 30569640
- [Background] Arnason TG, Bowen MW, Mansell KD. Effects of intermittent fasting on health markers in those with type 2 diabetes: A pilot study. World J Diabetes. 2017 Apr 15;8(4):154-164. doi: 10.4239/wjd.v8.i4.154. PMID 28465792
- [Background] Carter S, Clifton PM, Keogh JB. The effects of intermittent compared to continuous energy restriction on glycaemic control in type 2 diabetes; a pragmatic pilot trial. Diabetes Res Clin Pract. 2016 Dec;122:106-112. doi: 10.1016/j.diabres.2016.10.010. Epub 2016 Oct 19. PMID 27833048
- [Background] Harvie MN, Pegington M, Mattson MP, Frystyk J, Dillon B, Evans G, Cuzick J, Jebb SA, Martin B, Cutler RG, Son TG, Maudsley S, Carlson OD, Egan JM, Flyvbjerg A, Howell A. The effects of intermittent or continuous energy restriction on weight loss and metabolic disease risk markers: a randomized trial in young overweight women. Int J Obes (Lond). 2011 May;35(5):714-27. doi: 10.1038/ijo.2010.171. Epub 2010 Oct 5. PMID 20921964
- [Background] Jebeile H, Gow ML, Lister NB, Mosalman Haghighi M, Ayer J, Cowell CT, Baur LA, Garnett SP. Intermittent Energy Restriction Is a Feasible, Effective, and Acceptable Intervention to Treat Adolescents with Obesity. J Nutr. 2019 Jul 1;149(7):1189-1197. doi: 10.1093/jn/nxz049. PMID 31006807
- [Background] Gabel K, Varady KA. Current research: effect of time restricted eating on weight and cardiometabolic health. J Physiol. 2022 Mar;600(6):1313-1326. doi: 10.1113/JP280542. Epub 2020 Oct 21. PMID 33002219
- [Background] Chaix A, Manoogian ENC, Melkani GC, Panda S. Time-Restricted Eating to Prevent and Manage Chronic Metabolic Diseases. Annu Rev Nutr. 2019 Aug 21;39:291-315. doi: 10.1146/annurev-nutr-082018-124320. Epub 2019 Jun 10. PMID 31180809
- [Background] Martens CR, Rossman MJ, Mazzo MR, Jankowski LR, Nagy EE, Denman BA, Richey JJ, Johnson SA, Ziemba BP, Wang Y, Peterson CM, Chonchol M, Seals DR. Short-term time-restricted feeding is safe and feasible in non-obese healthy midlife and older adults. Geroscience. 2020 Apr;42(2):667-686. doi: 10.1007/s11357-020-00156-6. Epub 2020 Jan 23. PMID 31975053
- [Background] Vidmar AP, Goran MI, Raymond JK. Time-Limited Eating in Pediatric Patients with Obesity: A Case Series. J Food Sci Nutr Res. 2019;2(3):236-244. doi: 10.26502/jfsnr.2642-11000022. Epub 2019 Sep 20. PMID 32455345
- [Background] Cienfuegos S, Gabel K, Kalam F, Ezpeleta M, Wiseman E, Pavlou V, Lin S, Oliveira ML, Varady KA. Effects of 4- and 6-h Time-Restricted Feeding on Weight and Cardiometabolic Health: A Randomized Controlled Trial in Adults with Obesity. Cell Metab. 2020 Sep 1;32(3):366-378.e3. doi: 10.1016/j.cmet.2020.06.018. Epub 2020 Jul 15. PMID 32673591
- [Background] Gabel K, Hoddy KK, Haggerty N, Song J, Kroeger CM, Trepanowski JF, Panda S, Varady KA. Effects of 8-hour time restricted feeding on body weight and metabolic disease risk factors in obese adults: A pilot study. Nutr Healthy Aging. 2018 Jun 15;4(4):345-353. doi: 10.3233/NHA-170036. PMID 29951594
- [Background] Kesztyus D, Cermak P, Gulich M, Kesztyus T. Adherence to Time-Restricted Feeding and Impact on Abdominal Obesity in Primary Care Patients: Results of a Pilot Study in a Pre-Post Design. Nutrients. 2019 Nov 21;11(12):2854. doi: 10.3390/nu11122854. PMID 31766465
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Goodpaster BH, Sparks LM. Metabolic Flexibility in Health and Disease. Cell Metab. 2017 May 2;25(5):1027-1036. doi: 10.1016/j.cmet.2017.04.015. PMID 28467922
- [Background] Nogueira-de-Almeida CA, de Mello ED. Different Criteria for the Definition of Insulin Resistance and Its Relation with Dyslipidemia in Overweight and Obese Children and Adolescents. Pediatr Gastroenterol Hepatol Nutr. 2018 Jan;21(1):59-67. doi: 10.5223/pghn.2018.21.1.59. Epub 2018 Jan 12. PMID 29383306
- [Background] Gomez-Bruton A, Arenaza L, Medrano M, Mora-Gonzalez J, Cadenas-Sanchez C, Migueles JH, Munoz-Hernandez V, Merchan-Ramirez E, Martinez-Avila WD, Maldonado J, Oses M, Tobalina I, Gracia-Marco L, Vicente-Rodriguez G, Ortega FB, Labayen I. Associations of dietary energy density with body composition and cardiometabolic risk in children with overweight and obesity: role of energy density calculations, under-reporting energy intake and physical activity. Br J Nutr. 2019 May;121(9):1057-1068. doi: 10.1017/S0007114519000278. Epub 2019 Feb 6. PMID 30724143
- [Background] Wiegman A, Gidding SS, Watts GF, Chapman MJ, Ginsberg HN, Cuchel M, Ose L, Averna M, Boileau C, Boren J, Bruckert E, Catapano AL, Defesche JC, Descamps OS, Hegele RA, Hovingh GK, Humphries SE, Kovanen PT, Kuivenhoven JA, Masana L, Nordestgaard BG, Pajukanta P, Parhofer KG, Raal FJ, Ray KK, Santos RD, Stalenhoef AF, Steinhagen-Thiessen E, Stroes ES, Taskinen MR, Tybjaerg-Hansen A, Wiklund O; European Atherosclerosis Society Consensus Panel. Familial hypercholesterolaemia in children and adolescents: gaining decades of life by optimizing detection and treatment. Eur Heart J. 2015 Sep 21;36(36):2425-37. doi: 10.1093/eurheartj/ehv157. Epub 2015 May 25. PMID 26009596
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Background] Rueda Jaimes GE, Diaz Martinez LA, Ortiz Barajas DP, Pinzon Plata C, Rodriguez Martinez J, Cadena Afanador LP. [Validation of the SCOFF questionnaire for screening the eating behaviour disorders of adolescents in school]. Aten Primaria. 2005 Feb 15;35(2):89-94. doi: 10.1157/13071915. Spanish. PMID 15727751
- [Background] Vioque J, Navarrete-Munoz EM, Gimenez-Monzo D, Garcia-de-la-Hera M, Granado F, Young IS, Ramon R, Ballester F, Murcia M, Rebagliato M, Iniguez C; INMA-Valencia Cohort Study. Reproducibility and validity of a food frequency questionnaire among pregnant women in a Mediterranean area. Nutr J. 2013 Feb 19;12:26. doi: 10.1186/1475-2891-12-26. PMID 23421854
- [Background] Martinez-Gonzalez MA, Fernandez-Jarne E, Serrano-Martinez M, Marti A, Martinez JA, Martin-Moreno JM. Mediterranean diet and reduction in the risk of a first acute myocardial infarction: an operational healthy dietary score. Eur J Nutr. 2002 Aug;41(4):153-60. doi: 10.1007/s00394-002-0370-6. PMID 12242583
- [Background] Trichopoulou A, Costacou T, Bamia C, Trichopoulos D. Adherence to a Mediterranean diet and survival in a Greek population. N Engl J Med. 2003 Jun 26;348(26):2599-608. doi: 10.1056/NEJMoa025039. PMID 12826634
- [Background] Gerber M. Qualitative methods to evaluate Mediterranean diet in adults. Public Health Nutr. 2006 Feb;9(1A):147-51. doi: 10.1079/phn2005937. PMID 16512962
- [Background] Fung TT, Chiuve SE, McCullough ML, Rexrode KM, Logroscino G, Hu FB. Adherence to a DASH-style diet and risk of coronary heart disease and stroke in women. Arch Intern Med. 2008 Apr 14;168(7):713-20. doi: 10.1001/archinte.168.7.713. PMID 18413553
- [Background] Patterson RE, Haines PS, Popkin BM. Diet quality index: capturing a multidimensional behavior. J Am Diet Assoc. 1994 Jan;94(1):57-64. doi: 10.1016/0002-8223(94)92042-7. PMID 8270756
- [Background] Shivappa N, Steck SE, Hurley TG, Hussey JR, Hebert JR. Designing and developing a literature-derived, population-based dietary inflammatory index. Public Health Nutr. 2014 Aug;17(8):1689-96. doi: 10.1017/S1368980013002115. Epub 2013 Aug 14. PMID 23941862
- [Background] Marfell-Jones MJ, Stewart AD, de Ridder JH. International standards for anthropometric assessment. Wellington, New Zealand: International Society for the Advancement of Kinanthropometry. 2012.
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ. Recommendations for blood pressure measurement in humans and experimental animals: part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Circulation. 2005 Feb 8;111(5):697-716. doi: 10.1161/01.CIR.0000154900.76284.F6. PMID 15699287
- [Background] Cordero-MacIntyre ZR, Peters W, Libanati CR, Espana RC, Abila SO, Howell WH, Lohman TG. Reproducibility of DXA in obese women. J Clin Densitom. 2002 Spring;5(1):35-44. doi: 10.1385/jcd:5:1:035. PMID 11940727
- [Background] Gallagher D, Thornton JC, He Q, Wang J, Yu W, Bradstreet TE, Burke J, Heymsfield SB, Rivas VM, Kaufman R. Quantitative magnetic resonance fat measurements in humans correlate with established methods but are biased. Obesity (Silver Spring). 2010 Oct;18(10):2047-54. doi: 10.1038/oby.2010.97. Epub 2010 May 6. PMID 20448539
- [Background] Martinez-Nicolas A, Martinez-Madrid MJ, Almaida-Pagan PF, Bonmati-Carrion MA, Madrid JA, Rol MA. Assessing Chronotypes by Ambulatory Circadian Monitoring. Front Physiol. 2019 Nov 20;10:1396. doi: 10.3389/fphys.2019.01396. eCollection 2019. PMID 31824327
- [Background] Saint-Maurice PF, Welk GJ. Web-based assessments of physical activity in youth: considerations for design and scale calibration. J Med Internet Res. 2014 Dec 1;16(12):e269. doi: 10.2196/jmir.3626. PMID 25448192
- [Background] Ortega FB, Ruiz JR, Espana-Romero V, Vicente-Rodriguez G, Martinez-Gomez D, Manios Y, Beghin L, Molnar D, Widhalm K, Moreno LA, Sjostrom M, Castillo MJ; HELENA study group. The International Fitness Scale (IFIS): usefulness of self-reported fitness in youth. Int J Epidemiol. 2011 Jun;40(3):701-11. doi: 10.1093/ije/dyr039. Epub 2011 Mar 24. PMID 21441238
- [Background] Tomas Vila M, Miralles Torres A, Beseler Soto B. [Spanish version of the Pediatric Sleep Questionnaire (PSQ). A useful instrument in investigation of sleep disturbances in childhood. Reliability analysis]. An Pediatr (Barc). 2007 Feb;66(2):121-8. doi: 10.1157/13098928. Spanish. PMID 17306097
- [Background] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Background] Jauregui-Lobera I, Garcia-Cruz P, Carbonero-Carreno R, Magallares A, Ruiz-Prieto I. Psychometric properties of Spanish version of the Three-Factor Eating Questionnaire-R18 (Tfeq-Sp) and its relationship with some eating- and body image-related variables. Nutrients. 2014 Dec 4;6(12):5619-35. doi: 10.3390/nu6125619. PMID 25486370
- [Background] Dalton M, Finlayson G, Hill A, Blundell J. Preliminary validation and principal components analysis of the Control of Eating Questionnaire (CoEQ) for the experience of food craving. Eur J Clin Nutr. 2015 Dec;69(12):1313-7. doi: 10.1038/ejcn.2015.57. Epub 2015 Apr 8. PMID 25852028
- [Background] Banos RM, Cebolla A, Etchemendy E, Felipe S, Rasal P, Botella C. Validation of the Dutch Eating Behavior Questionnaire for Children (DEBQ-C) for use with Spanish children. Nutr Hosp. 2011 Jul-Aug;26(4):890-8. doi: 10.1590/S0212-16112011000400032. PMID 22470039
- [Background] Dalton M, Blundell J, Finlayson GS. Examination of food reward and energy intake under laboratory and free-living conditions in a trait binge eating subtype of obesity. Front Psychol. 2013 Oct 21;4:757. doi: 10.3389/fpsyg.2013.00757. eCollection 2013. PMID 24155732
- [Background] Epstein LH, Carr KA, Scheid JL, Gebre E, O'Brien A, Paluch RA, Temple JL. Taste and food reinforcement in non-overweight youth. Appetite. 2015 Aug;91:226-32. doi: 10.1016/j.appet.2015.04.050. Epub 2015 Apr 16. PMID 25891040
- [Background] Stevens K. Developing a descriptive system for a new preference-based measure of health-related quality of life for children. Qual Life Res. 2009 Oct;18(8):1105-13. doi: 10.1007/s11136-009-9524-9. Epub 2009 Aug 20. PMID 19693703
- [Background] Stevens K. Assessing the performance of a new generic measure of health-related quality of life for children and refining it for use in health state valuation. Appl Health Econ Health Policy. 2011 May 1;9(3):157-69. doi: 10.2165/11587350-000000000-00000. PMID 21506622
- [Background] Amaya-Arias AC, Alzate JP, Eslava-Schmalbach JH. Construct and Criterion Validity of the PedsQL 4.0 Instrument (Pediatric Quality of Life Inventory) in Colombia. Int J Prev Med. 2017 Aug 24;8:57. doi: 10.4103/ijpvm.IJPVM_194_16. eCollection 2017. PMID 28900536
- [Background] Wallander JL, Kerbawy S, Toomey S, Lowry R, Elliott MN, Escobar-Chaves SL, Franzini L, Schuster MA. Is obesity associated with reduced health-related quality of life in Latino, Black and White children in the community? Int J Obes (Lond). 2013 Jul;37(7):920-5. doi: 10.1038/ijo.2013.31. Epub 2013 Mar 12. PMID 23478424
- [Background] Revenga-Frauca J, Gonzalez-Gil EM, Bueno-Lozano G, De Miguel-Etayo P, Velasco-Martinez P, Rey-Lopez JP, Bueno-Lozano O, Moreno LA. Abdominal fat and metabolic risk in obese children and adolescents. J Physiol Biochem. 2009 Dec;65(4):415-20. doi: 10.1007/BF03185937. PMID 20358355
- [Background] Guil-Oumrait N, Valvi D, Garcia-Esteban R, Guxens M, Sunyer J, Torrent M, Casas M, Vrijheid M. Prenatal exposure to persistent organic pollutants and markers of obesity and cardiometabolic risk in Spanish adolescents. Environ Int. 2021 Jun;151:106469. doi: 10.1016/j.envint.2021.106469. Epub 2021 Mar 9. PMID 33711537
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Hoddy KK, Kroeger CM, Trepanowski JF, Barnosky AR, Bhutani S, Varady KA. Safety of alternate day fasting and effect on disordered eating behaviors. Nutr J. 2015 May 6;14:44. doi: 10.1186/s12937-015-0029-9. PMID 25943396
- See also: Related Info — http://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight